CLINICAL TRIAL: NCT01595685
Title: A Randomized, Open-label Trial Comparing Telbivudine vs, Entecavir in Reducing Serum HBsAg Levels in Patients With HBeAg-positive Chronic Hepatitis B Who Have Achieved Serum HBV DNA Undetectability by Preceding Entecavir Treatment
Brief Title: Telbivudine Versus Entecavir in Reducing Serum HBsAg Levels in Patients With HBeAg-positive Chronic Hepatitis B
Acronym: TERESA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Young-Suk Lim, Associate Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMC2012-0201
Record Dates: First submitted 2012-05-08; First posted 2012-05-10 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Viral Hepatitis B Without Delta-agent
Keywords: HBeAg-positive
MeSH Terms: interventions — Telbivudine; entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telbivudine (Experimental): Telbivudine 600 mg Daily Oral
  Interventions: Drug: Telbivudine
- Entecavir (Active Comparator): Entecavir 0.5 mg Daily Oral
  Interventions: Drug: Entecavir

INTERVENTIONS:
Drug: Telbivudine — Telbivudine 600 mg Daily Oral
  Other Names: Sebivo
  Arms: Telbivudine
Drug: Entecavir — Entecavir 0.5 mg Daily Oral
  Other Names: Baraclude
  Arms: Entecavir

SUMMARY:
The goal of chronic hepatitis B (CHB) treatment is complete and permanent eradication of hepatitis B virus (HBV) from patient's body, which is best represented by serum HBsAg loss accompanied by undetectable serum HBV DNA level.

While the most recently approved nucleos(t)ide analogues (NA) have marked antiviral potency and can induce HBV DNA undetectability in the majority of patients through prolonged treatment, NA need to be given long term, almost indefinitely, in most cases because they suppress HBV DNA only during therapy. For example, even after HBeAg-loss by a potent NA, suppression of serum HBV DNA to undetectable level is sustained only in about 23%-37% at 24 weeks off treatment. Thus, continuous therapy with NA until HBsAg clearance remains necessary in a majority of cases.

The recent availability of commercial quantitative assays of serum hepatitis B surface antigen (HBsAg) has enabled quantitative HBsAg to be used as a biomarker for prognosis and treatment response in CHB. It has been suggested that HBsAg decline during lamivudine or entecavir therapy is slower and less pronounced compared to interferon treatment, despite a higher effect on HBV DNA suppression. Based on HBsAg kinetics, it has been estimated that the predicted median time to HBsAg loss in patients treated with lamivudine or entecavir is more than 30 years. Thus, treatment that can induce rapid decline of HBsAg would have clear advantage in reducing the treatment duration required to achieve HBsAg-loss.

Interestingly, in a recent preliminary study, 24-weeks of treatment with telbivudine has induced HBsAg decline as comparable to pegylated interferon treatment. Although there has been no head-to-head trial comparing NAs in inducing HBsAg decline, previous studies consistently suggested that the decline of HBsAg is greater during telbivudine treatment compared with lamivudine or entecavir.

Thus, in this clinical trial, the investigators will investigate whether telbivudine is more effective in inducing HBsAg decline compared with entecavir in HBeAg-positive CHB patients who have achieved undetectable serum HBV DNA by preceding entecavir treatment.

DETAILED DESCRIPTION:
A single-center randomized active-controlled open-label superiority trial

* Patients will be randomly assigned 1:1 to receive telbivudine (600 mg/day) or ongoing entecavir (0.5 mg/day) for 48 weeks.
* Eligible patients will be randomized using blocks of permuted treatment assignments after stratification by HBsAg level (1,000 IU/mL-5,000 IU/mL and ≥5,000 IU/mL IU/mL) and by entecavir treatment duration (1 year-2 year, ≥2 year).
* Because over 98% of Korean patients with CHB have HBV genotype C,9 HBV genotype will not determined or be regarded as a stratification factor.
* There will be no interruption in entecavir therapy before randomization.
* Patients' treatment information will be retrospectively collected during entecavir treatment phase as well (DNA change, HBeAg status, HBsAg titre, ALT, and treatment duration. etc)
* Patients will be screened within 4 weeks before randomization to determine study eligibility.

ELIGIBILITY:
Inclusion Criteria: All of below

* HBsAg titer > 1,000 IU/mL
* HBeAg positive at study entry and at the baseline of ETV treatment
* HBV DNA undetectable (<15 IU/mL) at least 2 occasions of more than 3 months apart
* Treatment with entecavir (0.5 mg/day) for more than 1 year
* Patient is ambulatory.
* Patient is able and willing to give informed consent.

Exclusion Criteria: Any of below

* Prior exposure to oral nucloes(t)ide analogue other than entecavir
* Prior any exposure to interferon or pegylated interferon
* Cirrhosis with Child-Pugh score ≥8
* Hepatocellular carcinoma Identified or suspected
* Other malignancy
* Prior organ transplantation
* Under immunosuppressive agent
* Renal insufficiency (serum creatinine > 1.4)
* Pregnant woman or willing to be pregnant woman or man

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2012-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
HBsAg titer at 48 weeks | at 48 weeks

SECONDARY OUTCOMES:
Proportion of patients with serum HBsAg decline of ≥0.5 log10 IU/mL and <1.0 log10 IU/mL | at 48 weeks of treatment
Proportion of patients with serum HBsAg decline greater than 1.0 log10 IU/mL | at 48 weeks of treatment
Proportion of patients with serum HBsAg loss | at 48 weeks of treatment
Proportion of patients with serum HBeAg loss or HBeAg seroconversion | at 48 weeks of treatment
Proportion of patients with virologic rebound or genotypic resistance | up to 48 weeks of treatment
Proportion of patients with normal ALT | at 48 weeks of treatment
Adverse events: Creatine kinase level, GFR, Muscle events, Other AEs | up to 48 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Young-Suk Lim, M.D., Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] An J, Lim YS, Kim GA, Han SB, Jeong W, Lee D, Shim JH, Lee HC, Lee YS. Telbivudine versus entecavir in patients with undetectable hepatitis B virus DNA: a randomized trial. BMC Gastroenterol. 2017 Jan 19;17(1):15. doi: 10.1186/s12876-017-0572-2. PMID 28103819